CLINICAL TRIAL: NCT06677060
Title: A Phase III, Randomised, Placebo-controlled, Event-driven Study to Evaluate the Effect of Baxdrostat in Combination With Dapagliflozin Compared With Dapagliflozin Alone on the Risk of Incident Heart Failure and Cardiovascular Death
Brief Title: Phase III Study Investigating Heart Failure and Cardiovascular Death With Baxdrostat in Combination With Dapagliflozin
Acronym: Prevent-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D6973C00001; 2024-514506-32-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart failure: Baxdrostat; Dapagliflozin; cardiovascular
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baxdrostat/Dapagliflozin (Experimental): Participants randomised to the baxdrostat/dapagliflozin arm will initially receive a dose of baxdrostat lower dose and dapagliflozin. For participants that meet the up-titration criteria, baxdrostat may be up-titrated to higher dose.
  Interventions: Drug: Baxdrostat and dapagliflozin
- Placebo/Dapagliflozin (Experimental): Patients will receive a dose of dapagliflozin in combination with matching placebo
  Interventions: Other: Placebo and dapagliflozin

INTERVENTIONS:
Drug: Baxdrostat and dapagliflozin — baxdrostat tablet and dapagliflozin tablet
  Other Names: Baxdrostat CIN-107
  Arms: Baxdrostat/Dapagliflozin
Other: Placebo and dapagliflozin — placebo tablet and dapagliflozin tablet
  Arms: Placebo/Dapagliflozin

SUMMARY:
Participants include men and women ≥ 40 years of age with T2DM, established CV disease, a history of HTN with an SBP of at least 130 mmHg at screening, who meet the predefined serum potassium level, and with at least one additional risk factor for HF.

The study will include an optional pre-screening period to facilitate sites' identification of potentially eligible participants to enter the full screening assessments. Participants will not be required to visit the site and no informed consent is required for the optional pre-screening period. The pre-screening assessments do not replace the full screening tests at Visit 1.

Upon entering the screening period, all consented participants (after signature of screening ICF) will be screened during an up to 14-day screening period. Participants who meet all screening inclusion/exclusion criteria but are not treated with SGLT2i or are treated for less than 4 weeks will enter a run-in period with dapagliflozin 10 mg once daily for at least 4 weeks (and not more than 6 weeks) before randomisation.

Site visits will take place at approximately 2-, 4-, 8-, 16-, and 34-weeks following randomisation. Thereafter visits will occur approximately every 4 months.

The study closure procedures will be initiated when the predetermined number of the first secondary endpoint events (ie, the composite of hospitalisation for HF or CV death) is predicted to have occurred i.e., the PACD.

In case of premature discontinuation of the blinded study intervention, participants will remain in the study. Unless a participant meets the dapagliflozin specific discontinuation criteria, they will continue to receive open label dapagliflozin 10 mg. It is important that the scheduled study visits and data collection continue according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants of any sex and gender must be ≥ 40 years old at the time of signing the informed consent.
* Diagnosed with T2DM and requiring treatment
* Established CV disease (ischaemic heart disease, cerebrovascular disease, peripheral arterial disease)
* History of HTN and an SBP ≥ 130 mmHg at screening and ≥ 120 mmHg at the Randomisation Visit.
* At least one additional risk factor for HF:

  * Age ≥ 70 years
  * UACR > 20 mg/g
  * eGFR < 60 mL/min/1.73 m2
  * History of polyvascular disease (at least two of: ischaemic heart disease, cerebrovascular disease, and peripheral arterial disease)
  * History of atrial fibrillation or atrial flutter
  * NT-proBNP > 125 ng/L

Exclusion Criteria:

* Previously confirmed diagnosis and treatment of heart failure
* An eGFR < 30 mL/min/1.73 m2 at screening
* Known hyperkalaemia, defined as potassium ≥ 5.5 mmol/L within 3 months prior to screening
* Type 1 diabetes mellitus or uncontrolled T2DM with HbA1c > 10.5% (> 91 mmol/mol) at screening
* Serum sodium < 135 mmol/L at screening, determined as per central laboratory assessment
* Stroke, transient ischaemic cerebral attack, valve implantation or valve replacement, carotid surgery, carotid angioplasty, or cardiac surgery, within 3 months prior to randomisation
* Myocardial infarction within 3 months prior to randomisation, or within 1 month prior to randomisation when there is no further planned revascularisation
* Percutaneous coronary intervention within 1 month prior to randomisation
* Known severe hepatic impairment, defined as Child-Pugh Class C, based on records that confirm documented medical history
* Documented history of adrenal insufficiency
* Any dialysis (including for acute kidney injury) within 3 months prior to screening
* Any acute kidney injury within 3 months prior to screening
* Prohibited concomitant medications

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11300 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2029-12-17 (Estimated); Study Completion 2029-12-17 (Estimated)

PRIMARY OUTCOMES:
To determine if baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of an HF event or CV death | Event driven; Up to 38 months
  Time to first occurrence of any of the components of the composite of:
  * Hospitalisation for HF
  * HF without hospitalisation
  * CV death

SECONDARY OUTCOMES:
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of hospitalisation for HF or CV death | Event driven; Up to 38 months
  Time to first occurrence of any of the components of the composite of:
  * Hospitalisation for HF
  * CV death
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of HF events | Event driven; Up to 38 months
  Time to first occurrence of any of the components of the composite of:
  * Hospitalisation for HF
  * HF without hospitalisation
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of CV death | Event driven; Up to 38 months
  Time to CV death
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of all-cause mortality | Event driven; Up to 38 months
  Time to all-cause death
To determine whether baxdrostat/dapagliflozin is superior to placebo/dapagliflozin in reducing the risk of 4-point MACE (CV death, MI, stroke, and hospitalisation for HF) | Event driven; Up to 38 months
  Time to first occurrence of any of the components of the composite of:
  * CV death
  * MI
  * Stroke
  * Hospitalisation for HF

CONTACTS AND LOCATIONS:
Locations (715):
- United States (162):
  - Research Site, Birmingham, Alabama
  - Research Site, Centreville, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Vestavia Hills, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Dublin, California
  - Research Site, Huntington Beach, California
  - Research Site, Inglewood, California
  - Research Site, La Jolla, California
  - Research Site, Lakewood, California
  - Research Site, Lincoln, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, San Francisco, California
  - Research Site, Santa Maria, California
  - Research Site, Sherman Oaks, California
  - Research Site, Thousand Oaks, California
  - Research Site, Aurora, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Crystal River, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Albany, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Canton, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Cordele, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Island Lake, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Richmond, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, El Dorado, Kansas
  - Research Site, Lenexa, Kansas
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Beltsville, Maryland
  - Research Site, Lutherville-Timonium, Maryland
  - Research Site, Potomac, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, New Bedford, Massachusetts
  - Research Site, Roslindale, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Mankato, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Missoula, Montana
  - Research Site, Norfolk, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Carson City, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Pennington, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Massapequa, New York
  - Research Site, New York, New York
  - Research Site, Queens Village, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Kernersville, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Beavercreek, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Horsham, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Fort Mill, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Cleveland, Tennessee
  - Research Site, Morristown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Abilene, Texas
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Dallas, Texas
  - Research Site, Duncanville, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Mansfield, Texas
  - Research Site, McAllen, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Paris, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Stephenville, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tomball, Texas
  - Research Site, Weslaco, Texas
  - Research Site, Woodway, Texas
  - Research Site, Clearfield, Utah
  - Research Site, Roy, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Burke, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Redmond, Washington
  - Research Site, Renton, Washington
  - Research Site, Kingwood, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Green Bay, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Caba
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Nicolás
  - Research Site, San Nicolás de los Arroyos
  - Research Site, San Vicente
  - Research Site, Santa Fe
- Australia (13):
  - Research Site, Adelaide
  - Research Site, Elizabeth Vale
  - Research Site, Fremantle
  - Research Site, Geelong
  - Research Site, Kingswood
  - Research Site, Leabrook
  - Research Site, Maroubra
  - Research Site, Merewether
  - Research Site, Milton
  - Research Site, Mulgrave
  - Research Site, Osborne Park
  - Research Site, Rockhampton
  - Research Site, Wollongong
- Brazil (15):
  - Research Site, Belém
  - Research Site, Blumenau
  - Research Site, Bragança Paulista
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Juiz de Fora
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São José dos Campos
  - Research Site, São Paulo
  - Research Site, Tatuí
- Bulgaria (10):
  - Research Site, Haskovo
  - Research Site, Panagyurishte
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Canada (28):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Mirabel, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Regina, Saskatchewan
- China (46):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Heze
  - Research Site, Huangshi
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kaifeng
  - Research Site, Liaocheng
  - Research Site, Linhai
  - Research Site, Linyi
  - Research Site, Lishui
  - Research Site, Luoyang
  - Research Site, Meihekou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Nanyang
  - Research Site, Panjin
  - Research Site, Pingxiang
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Siping
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xianyang
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Zhumadian
  - Research Site, Zigong
- Czechia (14):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Broumov
  - Research Site, Chlumec nad Cidlinou
  - Research Site, Hodonín
  - Research Site, Humpolec
  - Research Site, Jílové u Prahy
  - Research Site, Krnov
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Police nad Metují
  - Research Site, Prague
- Denmark (17):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Aarhus N
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Frederiksberg
  - Research Site, Gistrup
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Hjørring
  - Research Site, Holbæk
  - Research Site, Hvidovre
  - Research Site, Roskilde
  - Research Site, Slagelse
  - Research Site, Svendborg
  - Research Site, Viborg
- France (27):
  - Research Site, Amiens
  - Research Site, Angers
  - Research Site, Aurillac
  - Research Site, Besançon
  - Research Site, Bobigny
  - Research Site, Bois-Guillaume
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, Clermont-Ferrand
  - Research Site, Colombes
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, Le Coudray
  - Research Site, Le Creusot
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villeurbanne
- Germany (49):
  - Research Site, Aachen
  - Research Site, Amberg
  - Research Site, Bad Homburg
  - Research Site, Bad Oeynhausen
  - Research Site, Bamberg
  - Research Site, Bechhofen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Brandenburg
  - Research Site, Bremen
  - Research Site, Cologne
  - Research Site, Deggingen
  - Research Site, Dresden
  - Research Site, Elsterwerda
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Friedrichsthal
  - Research Site, Fulda
  - Research Site, Gelnhausen
  - Research Site, Görlitz
  - Research Site, Hamburg
  - Research Site, Haßloch
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Kaiserslautern
  - Research Site, Kassel
  - Research Site, Langen
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Mannheim
  - Research Site, Markkleeberg
  - Research Site, Munich
  - Research Site, Münster
  - Research Site, Naunhof
  - Research Site, Neuruppin
  - Research Site, Nittendorf
  - Research Site, Obertshausen
  - Research Site, Oldenburg
  - Research Site, Osnabrück
  - Research Site, Papenburg
  - Research Site, Pirna
  - Research Site, Potsdam
  - Research Site, Reinfeld (Holstein)
  - Research Site, Völklingen
  - Research Site, Wallerfing
  - Research Site, Wangen
  - Research Site, Weinheim
  - Research Site, Zwenkau
- Greece (6):
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Hungary (14):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Kalocsa
  - Research Site, Nyíregyháza
  - Research Site, Nyíregyháza-Sóstóhegy
  - Research Site, Orosháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Szigetvár
  - Research Site, Szolnok
- India (16):
  - Research Site, Ahmedabad
  - Research Site, Ajmer
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Delhi
  - Research Site, Gūrgaon
  - Research Site, Hyderabad
  - Research Site, Kanpur
  - Research Site, Karamsad
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Secunderabad
  - Research Site, Surat
  - Research Site, Vijayawada
- Israel (9):
  - Research Site, Beersheba
  - Research Site, Be’er Ya‘aqov
  - Research Site, Haifa
  - Research Site, Herzelia
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (22):
  - Research Site, Alessandria
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Chiavari
  - Research Site, Cona
  - Research Site, Foggia
  - Research Site, Milan
  - Research Site, Mondovì
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Orbassano
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Potenza
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Rozzano
  - Research Site, Siena
  - Research Site, Torino
  - Research Site, Udine
- Japan (37):
  - Research Site, Amagasaki-shi
  - Research Site, Asahikawa-shi
  - Research Site, Azumino-shi
  - Research Site, Fukui-shi
  - Research Site, Hakusan-shi
  - Research Site, Himeji
  - Research Site, Itabashi-ku
  - Research Site, Izumo-shi
  - Research Site, Kakegawa-shi
  - Research Site, Kamakura-shi
  - Research Site, Kanazawa
  - Research Site, Kawaguchi-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kita-ku
  - Research Site, Kyoto
  - Research Site, Matsudo-shi
  - Research Site, Meguro-ku
  - Research Site, Mito
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Ogaki-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama-shi
  - Research Site, Sendai
  - Research Site, Shizuoka
  - Research Site, Suita-shi
  - Research Site, tabashi City
  - Research Site, Takamatsu
  - Research Site, Takatsuki-shi
  - Research Site, Toyota-Shi
  - Research Site, Tsuchiura-shi
  - Research Site, Ueda-shi
  - Research Site, Uwajima-shi
  - Research Site, Yanagawa-shi
  - Research Site, Yokkaichi-shi
  - Research Site, Yokohama
- Malaysia (11):
  - Research Site, Alor Star
  - Research Site, Johor Bahru
  - Research Site, Kota Samarahan
  - Research Site, Kuala Terengganu
  - Research Site, Kuantan
  - Research Site, Kuching
  - Research Site, Malacca
  - Research Site, Rawang
  - Research Site, Sarawak Miri
  - Research Site, Seri Manjung
  - Research Site, Sungai Buloh
- Mexico (14):
  - Research Site, Acapulco
  - Research Site, Aguascalientes
  - Research Site, Cuauhtémoc
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Monterrey
  - Research Site, Querétaro City
  - Research Site, San Juan del Río
  - Research Site, Veracruz
  - Research Site, Xalapa
  - Research Site, Zapopan
- Netherlands (15):
  - Research Site, 's-Hertogenbosch
  - Research Site, Almelo
  - Research Site, Amsterdam
  - Research Site, Born
  - Research Site, Deventer
  - Research Site, Ede
  - Research Site, Enschede
  - Research Site, Haarlem
  - Research Site, Harderwijk
  - Research Site, Hoogeveen
  - Research Site, Nijmegen
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Venlo
  - Research Site, Zwolle
- Peru (5):
  - Research Site, Bellavista
  - Research Site, Chorrillos
  - Research Site, Cusco
  - Research Site, Lima
  - Research Site, Piura
- Philippines (11):
  - Research Site, Angeles City
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Fuente Osmena Cebu City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Lipa City
  - Research Site, Manadaluyong City
  - Research Site, Puerto Princesa City
  - Research Site, Quezon City
  - Research Site, Roxas City
- Poland (29):
  - Research Site, Bialystok
  - Research Site, Biała Podlaska
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Chrzanów
  - Research Site, Częstochowa
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Jasło
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Myszków
  - Research Site, Olsztyn
  - Research Site, Ostrów Mazowiecka
  - Research Site, Piekary Śląskie
  - Research Site, Poznan
  - Research Site, Przemyśl
  - Research Site, Płock
  - Research Site, Radzionków
  - Research Site, Rzeszów
  - Research Site, Skórzewo
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Romania (9):
  - Research Site, Bacau
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Ploieşti
  - Research Site, Satu Mare
  - Research Site, Târgu Mureş
- Slovakia (14):
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Handlová
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Malacky
  - Research Site, Námestovo
  - Research Site, Prešov
  - Research Site, Prievidza
  - Research Site, Rimavská Sobota
  - Research Site, Rožňava
  - Research Site, Sabinov
  - Research Site, Svidník
- South Africa (19):
  - Research Site, Bellville
  - Research Site, Benoni
  - Research Site, Brackenfell
  - Research Site, Cape Town
  - Research Site, Centurion
  - Research Site, Claremont
  - Research Site, Diepkloof, Soweto
  - Research Site, Durban
  - Research Site, East London
  - Research Site, eMkhomazi
  - Research Site, Extension 8, Lenasia
  - Research Site, Lenasia
  - Research Site, Midrand
  - Research Site, Paarl
  - Research Site, Parow
  - Research Site, Pretoria
  - Research Site, Somerset West
  - Research Site, Wentworth
  - Research Site, Worcester
- South Korea (8):
  - Research Site, Bucheon-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju
  - Research Site, Yangsan
- Spain (11):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Sant Joan Despí
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vigo
- Sweden (8):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Huddinge
  - Research Site, Lund
  - Research Site, Mölndal
  - Research Site, Norrköping
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (9):
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (11):
  - Research Site, Bangkok
  - Research Site, Banphaeo
  - Research Site, Bansuan, Muang, Chonburi
  - Research Site, Chiang Mai
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Khlong Luang
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Naimuang
  - Research Site, Ubonratchathani
- Turkey (Türkiye) (13):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kahramanmaraş
  - Research Site, Kocaeli
  - Research Site, Kütahya
  - Research Site, Malatya
  - Research Site, Samsun
  - Research Site, Sivas
- Ukraine (7):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (17):
  - Research Site, Aberdeen
  - Research Site, Chesterfield
  - Research Site, Dundee
  - Research Site, Gatley
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Norwich
  - Research Site, Penzance
  - Research Site, Redruth
  - Research Site, Sandbach
  - Research Site, Southampton
  - Research Site, Stockton-on-Tees
  - Research Site, Swansea
  - Research Site, Weston-super-Mare
  - Research Site, Wolverhampton
  - Research Site, Woodbridge
  - Research Site, Yate
- Vietnam (7):
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Huế
  - Research Site, Rach Gia
  - Research Site, Vĩnh Yên

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/

REFERENCES:
- [Derived] Dwyer JP, Maklad N, Vedin O, Monyak J, Myte R, Chertow GM, Heerspink HJL, Little DJ. Efficacy and Safety of Baxdrostat in Participants with CKD and Uncontrolled Hypertension: A Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Sep 6. doi: 10.1681/ASN.0000000849. Online ahead of print. No abstract available. PMID 40913594